CLINICAL TRIAL: NCT01405196
Title: A Double-blind, Randomized, Placebo-controlled, Multicenter Dose-ranging Study To Evaluate The Efficacy And Safety Of Pf-04236921 In Subjects With Systemic Lupus Erythematosus (Sle)
Brief Title: Subcutaneous Treatment In Randomized Subjects To Evaluate Safety And Efficacy In Generalized Lupus Erythematosus
Acronym: BUTTERFLY
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B0151006; 2011-000420-15 (EudraCT Number); BUTTERFLY (Other: Alias Study Number)
Record Dates: First submitted 2011-07-27; First posted 2011-07-29 (Estimated); Results first posted 2017-12-19 (Actual); Last update posted 2017-12-19 (Actual); Status verified 2017-12

CONDITIONS: Lupus Erythematosus, Systemic
Keywords: double-blind; placebo-controlled; multicenter; dose-ranging; efficacy; safety; lupus.
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — PF-04236921

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 10 mg of PF-04236921 (Other)
  Interventions: Biological: PF-04236921
- 50 mg of PF-04236921 (Other)
  Interventions: Biological: PF-04236921
- 200 mg of PF-04236921 (Other)
  Interventions: Biological: PF-04236921
- Placebo (Other)
  Interventions: Biological: PF-04236921

INTERVENTIONS:
Biological: PF-04236921 — subcutaneous injection; administered at day 1, weeks 8, 16.
  Arms: 10 mg of PF-04236921
Biological: PF-04236921 — subcutaneous injection; administered at day 1, weeks 8, 16.
  Arms: 50 mg of PF-04236921
Biological: PF-04236921 — subcutaneous injection; administered at day 1, weeks 8, 16.
  Arms: 200 mg of PF-04236921
Biological: PF-04236921 — subcutaneous injection; administered at day 1, weeks 8, 16
  Arms: Placebo

SUMMARY:
The objective of this study is to evaluate and compare efficacy of 3 dose levels of PF-04236921 to placebo in subjects with generalized lupus using a measure called the Systemic Lupus Erythematosus (SLE) Responder Index. The study will evaluate secondary and exploratory measures as well.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects between ages of 18 and 75 years old at time of signing consent.
* Have a clinical diagnosis of SLE according to 1997 update on the revised 1982 American College of Rheumatology (ACR) criteria.
* Have a unequivocally positive anti-nuclear antibody (ANA) test result.
* Active disease at screening defined by both: SLEDAI-2K score greater than or equal to 6 and BILAG Level A disease in more than or equal to 1 organ system (except renal or central nervous system) or BILAG B disease in more than or equal to 2 organ systems if no level A disease in present.

Exclusion Criteria:

* Any prior history of treatment with PF-04236921, or anti-IL-6 agent;
* Have received any of the following within 364 days of day 1: a biologic investigational agent other than B cell targeted therapy; required 3 or more courses of systemic corticosteroids for concomitant conditions; history of previously untreated or current evidence of active or untreated latent infection with Tuberculosis (TB), evidence of prior untreated or currently active TB by chest radiography, residing with or frequent close contact with an individual with active TB.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2011-12 (Actual); Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (112):
- United States (67):
  - Anniston Medical Clinic, PC, Anniston, Alabama
  - Pinnacle Research Group, LLC, Anniston, Alabama
  - Achieve Clinical Research, LLC, Birmingham, Alabama
  - Med Investigations, Inc., Fair Oaks, California
  - Premier Clinical Research, LLC, Lakewood, California
  - Novo Research, Long Beach, California
  - St Mary Medical Center, Long Beach, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Wallace Rheumatic Study Center, Los Angeles, California
  - UCLA Division of Rheumatology, Los Angeles, California
  - UCLA Rheumatology Clinical Research Center, Los Angeles, California
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - UCLA Medical Center, Los Angeles, California
  - Inland Rheumatology and Osteoporosis Medical Group, Upland, California
  - Inland Rheumatology Clinical Trials, Inc., Upland, California
  - Asthma, Allergy, Arthritis and Lung Center, Daytona Beach, Florida
  - Southeastern Arthritis Center, Gainesville, Florida
  - Southeastern Community Pharmacy, Gainesville, Florida
  - Southeastern Integrated Medical, PL, d/b/a Florida Medical Research Institute, Gainesville, Florida
  - Southeastern lmaging & Diagnostics, Gainesville, Florida
  - New Horizon Research Center, Miami, Florida
  - Arthritis Associates, Orlando, Florida
  - Millennium Research, Ormond Beach, Florida
  - The Arthritis Center, Palm Harbor, Florida
  - Advent Clinical Research Centers, Inc., Pinellas Park, Florida
  - Burnette & Silverfield, MDS PLC, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Grady Health Systems, Atlanta, Georgia
  - Idaho Arthritis Center, Meridian, Idaho
  - University of Chicago Medical Center, Chicago, Illinois
  - Beacon Medical Group Rheumatology, Granger, Indiana
  - Indiana CTSI Clinical Research Center, Indianapolis, Indiana
  - Investigational Drug Services, Indianapolis, Indiana
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Johns Hopkins Outpatient Center, Baltimore, Maryland
  - Johns Hopkins Outpatient Express Testing Center, Baltimore, Maryland
  - Tufts Medical Center/ Center for Arthritis and Rheumatic Diseases, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - University of Michigan Health System, Ann Arbor, Michigan
  - University of Michigan Health System,, Ann Arbor, Michigan
  - Henry Ford Health System (Henry Ford Medical Center), Detroit, Michigan
  - Shores Rheumatology P.C, Saint Clair Shores, Michigan
  - University of Nevada School of Medicine, Las Vegas, Nevada
  - Albuquerque Clinical Trials, Albuquerque, New Mexico
  - Arthritis and Osteoporosis Medical Associates, PLLC, Brooklyn, New York
  - Feinstein Institute for Medical Research, Manhasset, New York
  - NYU Center for Musculoskeletal Care, New York, New York
  - Allergy/Immunology and Rheumatology, Rochester, New York
  - The University of North Carolina Clinical and Translational Research Center, Chapel Hill, North Carolina
  - The University of North Carolina Hospitals Investigational Drug Services, Chapel Hill, North Carolina
  - The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Joint and Muscle Medical Care, Charlotte, North Carolina
  - Box Arthritis & Rheumatology of the Carolinas, PLLC, Charlotte, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Paramount Medical Research and Consulting, LLC, Middleburg Heights, Ohio
  - Oklahoma Medical Research Foundation, Oklahoma City, Oklahoma
  - Clinical Research Center of Reading, LLP, Wyomissing, Pennsylvania
  - Low Country Rheumatology, PA/Low Country Research, Charleston, South Carolina
  - Arthritis Clinic, Jackson, Tennessee
  - West Tennessee Research Institute, Jackson, Tennessee
  - UT Southwestern Medical Center, Dallas, Texas
  - Rheumatic Disease Clinical Research Center, LLC, Houston, Texas
  - Accurate Clinical Research, Inc., Houston, Texas
  - Southwest Rheumatology Research, LLC, Mesquite, Texas
  - The Seattle Arthritis Clinic, Seattle, Washington
  - Tacoma Center for Arthritis Research, PS, Tacoma, Washington
  - Mountain State Clinical Research, Clarksburg, West Virginia
- Argentina (5):
  - Framingham Centro Medico, La Plata, Buenos Aires
  - Instituto CAICI S.R.L., Rosario, Santa Fe Province
  - Centro Medico Privado de Reumatologia, San Miguel de Tucumán, Tucumán Province
  - Centro de Educación Medica e Investigaciones Clinicas "Norberto Quirno" CEMIC, C.a.b.a
  - Centro Polivalente de Asistencia e Investigación Clínica - CER- San Juan, San Juan
- Chile (3):
  - Centro de Estudios Reumatologicos, Santiago, RM
  - Centro Medico Prosalud, Santiago, RM
  - Sociedad Medica del Aparato Locomotor S.A. (SOMEAL), Santiago, Santiago Metropolitan
- Colombia (11):
  - Centro Integral de Reumatologia REUMALAB S.A.S., Envigado, Antioquia
  - Hospital Pablo Tobon Uribe, Medellín, Antioquia
  - Mix Supplier S.A., Envigado, Antioquia, Colombia
  - Centro Integral de Reumatología del Caribe CIRCARIBE SAS, Barranquilla, Atlántico
  - Congregacion de Hermanas Franciscanas Misioneras de Maria Auxiliadora- Clinica Asunción, Barranquilla, Atlántico
  - Organizacion Clinica General del Norte S.A., Barranquilla, Atlántico
  - Farmamix Ltda., Bogota, Distrito Capital, Cundimarca
  - Centro Integral de Reumatologia e Inmunologia S.A.S.- CIREI S.A.S., Bogota, Cundinamarca
  - Riesgo De Fractura S.A, Bogota, Cundinamarca
  - Servimed E.U, Bucaramanga, Santander Department
  - Farmamix Ltda., Bogotá
- Germany (6):
  - Charité - Universitaetsmedizin Berlin, Berlin
  - Charité University Medicine Berlin. Schlosspark-Klinik, Berlin
  - Universitaetsklinikum Koeln, Cologne
  - Universitaetsklinikum Erlangen, Erlangen
  - CIRI am Klinikum der Goethe-Universitaet, Frankfurt am Main
  - Universitaetsklinikum Leipzig AoeR, Department fuer Innere Medizin, Leipzig
- Hungary (3):
  - Qualiclinic Kft., Budapest
  - Debreceni Egyetem Orvos és Egeszsegtudomanyi Centrum, Debrecen
  - Bekes Megyei Kepviselo-testulet Pandy Kalman Korhaz Infektologia, Hepatologia es Immunologia, Gyula
- Spitalul Clinic Republican, Chisinau, Md-2025, Moldova
- Peru (4):
  - Centro de Investigacion REUMED, Clinica Anglo Americana, San Isidro, Lima region
  - Investigaciones Clínicas SAC, Santiago de Surco, Lima region
  - Investigaciones Clinicas SAC, Surco, Lima region
  - Unidad de Investigación en Medicina Interna y Enfermedades Críticas, Arequipa
- Poland (4):
  - NZOZ Centrum Reumatologiczne Indywidualna Specjalistyczna Praktyka Lekarska lek.med. Barbara Bazela, Elblag
  - Medyczne Centrum Hetmanska - Indywidualna Specjalistyczna Praktyka Lekarska -, Poznan
  - Prywatna Praktyka Lekarska Prof. UM Dr hab. med. Pawel Hrycaj, Poznan
  - Centralny Szpital Kliniczny Ministerstwa Spraw Wewnetrznych, Warsaw
- Puerto Rico (2):
  - University of Puerto Rico, Rio Piedras
  - Division of Rheumatology, Allergy and Immunology, San Juan
- Romania (4):
  - Spitalul Clinic Sf. Maria, Bucharest
  - Spitalul Clinic Colentina, Bucharest
  - Spitalul Clinic Jedetean de urgenta Cluj, Reumatologie, Cluj-Napoca
  - Spitalul Clinic Judetean de Urgenta "Sf. Apostol Andrei", Galati
- Dong-A University Medical Center 1, Busan, South Korea
- National Taiwan University Hospital, Taipei TOC, Taiwan

REFERENCES:
- [Derived] Li C, Shoji S, Beebe J. Pharmacokinetics and C-reactive protein modelling of anti-interleukin-6 antibody (PF-04236921) in healthy volunteers and patients with autoimmune disease. Br J Clin Pharmacol. 2018 Sep;84(9):2059-2074. doi: 10.1111/bcp.13641. Epub 2018 Jun 25. PMID 29776017
- [Derived] Wallace DJ, Strand V, Merrill JT, Popa S, Spindler AJ, Eimon A, Petri M, Smolen JS, Wajdula J, Christensen J, Li C, Diehl A, Vincent MS, Beebe J, Healey P, Sridharan S. Efficacy and safety of an interleukin 6 monoclonal antibody for the treatment of systemic lupus erythematosus: a phase II dose-ranging randomised controlled trial. Ann Rheum Dis. 2017 Mar;76(3):534-542. doi: 10.1136/annrheumdis-2016-209668. Epub 2016 Sep 26. PMID 27672124
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B0151006&StudyName=Subcutaneous%20Treatment%20In%20Randomized%20Subjects%20To%20Evaluate%20Safety%20And%20Efficacy%20In%20Generalized%20Lupus%20Erythematosus%0A%20%20

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Due to safety reason, dosing in 200 mg reporting arm was prematurely terminated and the participants were discontinued from it. Therefore, the statistical analysis plan was amended after it and 200 mg reporting arm was not included in efficacy data analysis.
Groups:
- PF-04236921 10 Milligram (10 mg): Participants received 10 mg dose of PF-04236921 subcutaneously in the anterolateral right and left thighs at Week 0, Week 8 and Week 16.
- PF-04236921 50 mg: Participants received 50 mg dose of PF-04236921 subcutaneously in the anterolateral right and left thighs at Week 0, Week 8 and Week 16.
- PF-04236921 200 mg: Participants received 200 mg dose of PF-04236921 subcutaneously in the anterolateral right and left thighs at Week 0, Week 8 and Week 16.
- Placebo: Placebo matching to PF-04236921 administered subcutaneously in the anterolateral right and left thighs at Week 0, Week 8 and Week 16.
Period: Overall Study
Arm/Group | PF-04236921 10 Milligram (10 mg) | PF-04236921 50 mg | PF-04236921 200 mg | Placebo
Started | 45 | 47 | 46 | 45
Completed | 34 | 35 | 23 | 36
Not Completed | 11 | 12 | 23 | 9
Not completed — Study Terminated by Sponsor | 0 | 0 | 9 | 0
Not completed — Other | 2 | 2 | 5 | 0
Not completed — Withdrawal by Subject | 4 | 6 | 3 | 6
Not completed — Adverse Event | 2 | 2 | 0 | 2
Not completed — Death | 1 | 0 | 3 | 0
Not completed — Lost to Follow-up | 2 | 2 | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PF-04236921 10 Milligram (10 mg) | PF-04236921 50 mg | PF-04236921 200 mg | Placebo | Total
Number analyzed (Participants) | 45 | 47 | 46 | 45 | 183
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.9 (11.48) | 38.3 (10.49) | 41.3 (11.29) | 42.3 (13.04) | 40.4 (11.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 44 | 43 | 38 | 168
  Male | 2 | 3 | 3 | 7 | 15

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Systemic Lupus Erythematosus (SLE) Responder Index (SRI) at Week 24
Description: SRI components include:Systemic Lupus Erythematosus Disease Activity Index 2000(SLEDAI-2K),British Isles Lupus Assessment Group(BILAG) 2004,Physician's Global Assessment(PhGA).Participants classified as responder if they did not meet definition of treatment failure and met all the following criteria: greater than or equal to(>=) 4 point reduction in SLEDAI-2K score; no new BILAG A organ domain score or 2 new BILAG B organ domain scores; no worsening (less than [<] 0.3 point increase) in PhGA score. Treatment failure: any new/increased use of corticosteroids,immunosuppressants/antimalarial drug, any death, hospitalization/treatment discontinuation due to SLE, any flare of lupus interfering with participation in study. SLEDAI-2K:assesses improvement in disease activity (range: 0 to 105; higher score = higher severity). BILAG:assesses disease extent, severity (range: A[severe] to E[no disease]). PhGA: assesses worsening in participant's general health status(range: 0[none] to 3[severe]).
Time Frame: Week 24
Population: Full Analysis Set= all randomized participants who received at least 1 dose of study drug. Number of participants analyzed= participants who completed through the Week 24 visit. As per sponsor's decision, dosing in "PF-04236921 200 mg" arm was prematurely terminated and hence it was not included in efficacy analysis.
Measure: Number; unit: Percentage of participants
Arm/Group | PF-04236921 10 Milligram (10 mg) | PF-04236921 50 mg | Placebo
Number analyzed (Participants) | 35 | 36 | 42
Percentage of participants | 59.9 | 39.2 | 40.1
Statistical Analysis 1: Comparison: PF-04236921 10 Milligram (10 mg) vs Placebo; Point estimates of the Odds ratio (ORs) as well as their confidence intervals were calculated from the generalized linear mix model that included fixed factors of the stratification factors, treatment, visit and treatment by visit; Test type: Superiority; p = 0.076, Mixed Models Analysis — P-value was displayed without adjusting for multiplicity; Odds Ratio (OR) = 2.23, 90% CI 2-sided [0.89 to 5.62]
Statistical Analysis 2: Comparison: PF-04236921 50 mg vs Placebo; Point estimates of the ORs as well as their confidence intervals were calculated from the generalized linear mix model that included fixed factors of the stratification factors, treatment, visit and treatment by visit; Test type: Superiority; p = 0.528, Mixed Models Analysis — P-value was displayed without adjusting for multiplicity; Odds Ratio (OR) = 0.96, 90% CI 2-sided [0.38 to 2.41]

2. Secondary Outcome: Percentage of Participants Achieving Systemic Lupus Erythematosus (SLE) Responder Index (SRI) at Week 4, 8, 12, 16, and 20
Description: SRI components include:SLEDAI-2K ,BILAG 2004, PhGA. Participants classified as responder if they did not meet definition of treatment failure and met all the following criteria: >=4 point reduction in SLEDAI-2K score; no new BILAG A organ domain score or 2 new BILAG B organ domain scores; no worsening (<0.3 point increase) in PhGA score. Treatment failure: any new/increased use of corticosteroids,immunosuppressants/antimalarial drug, any death, hospitalization/treatment discontinuation due to SLE, any flare of lupus interfering with participation in study. SLEDAI-2K: assesses improvement in disease activity (range: 0 to 105; higher score = higher severity). BILAG:assesses disease extent, severity (range: A [severe] to E [no disease]). PhGA: assesses worsening in participant's general health status(range: 0[none] to 3[severe]).
Time Frame: Week 4, 8, 12, 16, 20
Population: Full Analysis Set= all randomized participants who received at least 1 dose of study drug. Here, "number analyzed" signifies those participants who were evaluable at specified time points. As per sponsor's decision, dosing in "PF-04236921 200 mg" arm was prematurely terminated and hence it was not included in efficacy analysis.
Measure: Number; unit: Percentage of participants
Arm/Group | PF-04236921 10 Milligram (10 mg) | PF-04236921 50 mg | Placebo
Number analyzed (Participants) | 45 | 47 | 45
Percentage of participants
  Week 4: number analyzed (Participants) | 43 | 44 | 45
  Week 4 | 12.2 | 7.1 | 4.8
  Week 8: number analyzed (Participants) | 43 | 43 | 43
  Week 8 | 26.8 | 21.5 | 26.3
  Week 12: number analyzed (Participants) | 39 | 41 | 42
  Week 12 | 33.7 | 20 | 36.3
  Week 16: number analyzed (Participants) | 36 | 39 | 41
  Week 16 | 48.9 | 28.9 | 37.1
  Week 20: number analyzed (Participants) | 36 | 39 | 43
  Week 20 | 54.7 | 36.8 | 38.3
Statistical Analysis 1: Comparison: PF-04236921 10 Milligram (10 mg) vs Placebo; Week 4: Point estimates of the ORs as well as their confidence intervals were calculated from the generalized linear mix model that included fixed factors of the stratification factors, treatment, visit and treatment by visit; Test type: Superiority; Odds Ratio (OR) = 2.77, 90% CI 2-sided [0.62 to 12.40]
Statistical Analysis 2: Comparison: PF-04236921 50 mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; Odds Ratio (OR) = 1.54, 90% CI 2-sided [0.31 to 7.71]
Statistical Analysis 3: Comparison: PF-04236921 10 Milligram (10 mg) vs Placebo; Week 8: Point estimates of the ORs as well as their confidence intervals were calculated from the generalized linear mix model that included fixed factors of the stratification factors, treatment, visit and treatment by visit; Test type: Superiority; Odds Ratio (OR) = 1.03, 90% CI 2-sided [0.40 to 2.67]
Statistical Analysis 4: Comparison: PF-04236921 50 mg vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority; Odds Ratio (OR) = 0.77, 90% CI 2-sided [0.29 to 2.05]
Statistical Analysis 5: Comparison: PF-04236921 10 Milligram (10 mg) vs Placebo; Week 12: Point estimates of the ORs as well as their confidence intervals were calculated from the generalized linear mix model that included fixed factors of the stratification factors, treatment, visit and treatment by visit; Test type: Superiority; Odds Ratio (OR) = 0.89, 90% CI 2-sided [0.35 to 2.24]
Statistical Analysis 6: Comparison: PF-04236921 50 mg vs Placebo; [analysis description as in outcome 2, analysis 5]; Test type: Superiority; Odds Ratio (OR) = 0.44, 90% CI 2-sided [0.16 to 1.16]
Statistical Analysis 7: Comparison: PF-04236921 10 Milligram (10 mg) vs Placebo; Week 16: Point estimates of the ORs as well as their confidence intervals were calculated from the generalized linear mix model that included fixed factors of the stratification factors, treatment, visit and treatment by visit; Test type: Superiority; Odds Ratio (OR) = 1.62, 90% CI 2-sided [0.64 to 4.09]
Statistical Analysis 8: Comparison: PF-04236921 50 mg vs Placebo; [analysis description as in outcome 2, analysis 7]; Test type: Superiority; Odds Ratio (OR) = 0.69, 90% CI 2-sided [0.27 to 1.77]
Statistical Analysis 9: Comparison: PF-04236921 10 Milligram (10 mg) vs Placebo; Week 20: Point estimates of the ORs as well as their confidence intervals were calculated from the generalized linear mix model that included fixed factors of the stratification factors, treatment, visit and treatment by visit; Test type: Superiority; Odds Ratio (OR) = 1.95, 90% CI 2-sided [0.78 to 4.84]
Statistical Analysis 10: Comparison: PF-04236921 50 mg vs Placebo; [analysis description as in outcome 2, analysis 9]; Test type: Superiority; Odds Ratio (OR) = 0.94, 90% CI 2-sided [0.38 to 2.32]

3. Secondary Outcome: Percentage of Participants Achieving Modified Systemic Lupus Erythematosus (SLE) Responder Index (SRI) at Week 4, 8, 12, 16, 20, and 24
Description: SRI components include: modified SLEDAI-2K (SLEDAI-2K without standard parameters "Low complement" and "Leukopenia"), BILAG 2004, PhGA. Participants classified as responder if they did not meet definition of treatment failure and met all the following criteria: >=4 point reduction in SLEDAI-2K score; no new BILAG A organ domain score or 2 new BILAG B organ domain scores; no worsening (<0.3 point increase) in PhGA score. Treatment failure: any new/increased use of corticosteroids, immunosuppressants/antimalarial drug, any death, hospitalization/treatment discontinuation due to SLE, any flare of lupus interfering with participation in study. Modified SLEDAI-2K: assesses improvement in disease activity (range: 0 to 102; higher score = higher severity). BILAG: assesses disease extent, severity (range: A [severe] to E [no disease]). PhGA: assesses worsening in participant's general health status (range: 0[none] to 3[severe]).
Time Frame: Week 4, 8, 12, 16, 20, 24
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | PF-04236921 10 Milligram (10 mg) | PF-04236921 50 mg | Placebo
Number analyzed (Participants) | 45 | 47 | 45
Percentage of participants
  Week 4: number analyzed (Participants) | 43 | 44 | 45
  Week 4 | 9.5 | 7 | 9.2
  Week 8: number analyzed (Participants) | 43 | 43 | 43
  Week 8 | 23.8 | 25.7 | 30.2
  Week 12: number analyzed (Participants) | 39 | 41 | 42
  Week 12 | 35.6 | 24.9 | 42.6
  Week 16: number analyzed (Participants) | 36 | 39 | 41
  Week 16 | 50.2 | 34 | 41
  Week 20: number analyzed (Participants) | 36 | 39 | 43
  Week 20 | 56.5 | 46.9 | 42.2
  Week 24: number analyzed (Participants) | 35 | 36 | 42
  Week 24 | 61.2 | 41.4 | 41.6
Statistical Analysis 1: Comparison: PF-04236921 10 Milligram (10 mg) vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; Odds Ratio (OR) = 1.05, 90% CI 2-sided [0.28 to 3.88]
Statistical Analysis 2: Comparison: PF-04236921 50 mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; Odds Ratio (OR) = 0.75, 90% CI 2-sided [0.19 to 3.01]
Statistical Analysis 3: Comparison: PF-04236921 10 Milligram (10 mg) vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority; Odds Ratio (OR) = 0.72, 90% CI 2-sided [0.28 to 1.85]
Statistical Analysis 4: Comparison: PF-04236921 50 mg vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority; Odds Ratio (OR) = 0.80, 90% CI 2-sided [0.32 to 2.02]
Statistical Analysis 5: Comparison: PF-04236921 10 Milligram (10 mg) vs Placebo; [analysis description as in outcome 2, analysis 5]; Test type: Superiority; Odds Ratio (OR) = 0.75, 90% CI 2-sided [0.30 to 1.83]
Statistical Analysis 6: Comparison: PF-04236921 50 mg vs Placebo; [analysis description as in outcome 2, analysis 5]; Test type: Superiority; Odds Ratio (OR) = 0.45, 90% CI 2-sided [0.18 to 1.13]
Statistical Analysis 7: Comparison: PF-04236921 10 Milligram (10 mg) vs Placebo; [analysis description as in outcome 2, analysis 7]; Test type: Superiority; Odds Ratio (OR) = 1.45, 90% CI 2-sided [0.58 to 3.60]
Statistical Analysis 8: Comparison: PF-04236921 50 mg vs Placebo; [analysis description as in outcome 2, analysis 7]; Test type: Superiority; Odds Ratio (OR) = 0.74, 90% CI 2-sided [0.30 to 1.84]
Statistical Analysis 9: Comparison: PF-04236921 10 Milligram (10 mg) vs Placebo; [analysis description as in outcome 2, analysis 9]; Test type: Superiority; Odds Ratio (OR) = 1.78, 90% CI 2-sided [0.72 to 4.37]
Statistical Analysis 10: Comparison: PF-04236921 50 mg vs Placebo; [analysis description as in outcome 2, analysis 9]; Test type: Superiority; Odds Ratio (OR) = 1.21, 90% CI 2-sided [0.50 to 2.92]
Statistical Analysis 11: Comparison: PF-04236921 10 Milligram (10 mg) vs Placebo; Week 24: Point estimates of the ORs as well as their confidence intervals were calculated from the generalized linear mix model that included fixed factors of the stratification factors, treatment, visit and treatment by visit; Test type: Superiority; Odds Ratio (OR) = 2.22, 90% CI 2-sided [0.89 to 5.55]
Statistical Analysis 12: Comparison: PF-04236921 50 mg vs Placebo; [analysis description as in outcome 3, analysis 11]; Test type: Superiority; Odds Ratio (OR) = 1.00, 90% CI 2-sided [0.40 to 2.46]

4. Secondary Outcome: Percentage of Participants Achieving British Isles Lupus Assessment Group-based Composite Lupus Assessment (BICLA) Response at Week 4, 8, 12, 16, 20, and 24
Description: BICLA include: BILAG-2004, SLEDAI-2K, PhGA of disease activity. Participants classified as responder if they did not meet the definition of treatment failure and met all the following criteria: BILAG-2004 improvement (all A scores at baseline improved to B/C/D and all B scores improved to C or D); no worsening in disease activity (no new BILAG-2004 A scores or =<1 new B score); no worsening of total SLEDAI-2K score; no significant deterioration (<10 percent [%] worsening) in analogue PhGA. Treatment failure: any new/increased use of corticosteroids,immunosuppressants/antimalarial, any death, hospitalization/treatment discontinuation due to SLE, any flare of lupus interfering with participation in study. BILAG:assesses disease extent, severity (range: A[severe] to E[no disease]). SLEDAI-2K:assesses improvement in disease activity (range: 0 to 105; higher score = higher severity). PhGA: assesses worsening in participant's general health status(range: 0[none] to 3[severe]).
Time Frame: Week 4, 8, 12, 16, 20, 24
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | PF-04236921 10 Milligram (10 mg) | PF-04236921 50 mg | Placebo
Number analyzed (Participants) | 45 | 47 | 45
Percentage of participants
  Week 4: number analyzed (Participants) | 43 | 44 | 45
  Week 4 | 26.2 | 21.7 | 21
  Week 8: number analyzed (Participants) | 43 | 43 | 43
  Week 8 | 26.2 | 29 | 30.6
  Week 12: number analyzed (Participants) | 39 | 41 | 42
  Week 12 | 33.6 | 39.6 | 33.3
  Week 16: number analyzed (Participants) | 36 | 39 | 41
  Week 16 | 45.5 | 39.2 | 26.2
  Week 20: number analyzed (Participants) | 35 | 39 | 43
  Week 20 | 43.7 | 31.6 | 21.7
  Week 24: number analyzed (Participants) | 35 | 36 | 42
  Week 24 | 49.7 | 40.5 | 25.1
Statistical Analysis 1: Comparison: PF-04236921 10 Milligram (10 mg) vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; Odds Ratio (OR) = 1.34, 90% CI 2-sided [0.53 to 3.35]
Statistical Analysis 2: Comparison: PF-04236921 50 mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; Odds Ratio (OR) = 1.04, 90% CI 2-sided [0.41 to 2.65]
Statistical Analysis 3: Comparison: PF-04236921 10 Milligram (10 mg) vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority; Odds Ratio (OR) = 0.81, 90% CI 2-sided [0.33 to 1.96]
Statistical Analysis 4: Comparison: PF-04236921 50 mg vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority; Odds Ratio (OR) = 0.93, 90% CI 2-sided [0.39 to 2.23]
Statistical Analysis 5: Comparison: PF-04236921 10 Milligram (10 mg) vs Placebo; [analysis description as in outcome 2, analysis 5]; Test type: Superiority; Odds Ratio (OR) = 1.01, 90% CI 2-sided [0.42 to 2.45]
Statistical Analysis 6: Comparison: PF-04236921 50 mg vs Placebo; [analysis description as in outcome 2, analysis 5]; Test type: Superiority; Odds Ratio (OR) = 1.31, 90% CI 2-sided [0.55 to 3.10]
Statistical Analysis 7: Comparison: PF-04236921 10 Milligram (10 mg) vs Placebo; [analysis description as in outcome 2, analysis 7]; Test type: Superiority; Odds Ratio (OR) = 2.36, 90% CI 2-sided [0.95 to 5.88]
Statistical Analysis 8: Comparison: PF-04236921 50 mg vs Placebo; [analysis description as in outcome 2, analysis 7]; Test type: Superiority; Odds Ratio (OR) = 1.82, 90% CI 2-sided [0.74 to 4.46]
Statistical Analysis 9: Comparison: PF-04236921 10 Milligram (10 mg) vs Placebo; [analysis description as in outcome 2, analysis 9]; Test type: Superiority; Odds Ratio (OR) = 2.80, 90% CI 2-sided [1.10 to 7.12]
Statistical Analysis 10: Comparison: PF-04236921 50 mg vs Placebo; [analysis description as in outcome 2, analysis 9]; Test type: Superiority; Odds Ratio (OR) = 1.67, 90% CI 2-sided [0.66 to 4.21]
Statistical Analysis 11: Comparison: PF-04236921 10 Milligram (10 mg) vs Placebo; [analysis description as in outcome 3, analysis 11]; Test type: Superiority; Odds Ratio (OR) = 2.95, 90% CI 2-sided [1.18 to 7.41]
Statistical Analysis 12: Comparison: PF-04236921 50 mg vs Placebo; [analysis description as in outcome 3, analysis 11]; Test type: Superiority; Odds Ratio (OR) = 2.03, 90% CI 2-sided [0.82 to 5.06]

5. Secondary Outcome: Percentage of Participants Achieving Pre-defined Criteria for Systemic Lupus Erythematosus (SLE) Responder Index (SRI) Components at Week 24
Description: SRI components include: SLEDAI-2K, BILAG 2004 and PhGA. Participants classified as responder if they did not meet definition of treatment failure and met all the following criteria: >=4 point reduction in SLEDAI-2K score; no new BILAG A organ domain score or 2 new BILAG B organ domain scores; no worsening(<0.3 point increase) in PhGA score. Treatment failure: any new/increased use of corticosteroids, immunosuppressants/antimalarial drug, any death, hospitalization/treatment discontinuation due to SLE, any flare of lupus interfering with participation in study. SLEDAI-2K: assesses improvement in disease activity(range: 0 to 105; higher score = higher severity). BILAG: assesses disease extent, severity (range: A[severe] to E [no disease]). PhGA: assesses worsening in participant's general health status (range: 0[none] to 3[severe]). Model percent estimates reported only for 'Reduction in SLEDAI Score','No Worsening in PhGA' categories; for remaining categories, raw percentages reported
Time Frame: Week 24
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | PF-04236921 10 Milligram (10 mg) | PF-04236921 50 mg | Placebo
Number analyzed (Participants) | 34 | 36 | 41
Percentage of participants
  4 or More Points Reduction in SLEDAI Score | 60.7 | 44.9 | 49.3
  No New 1A/2B BILAG | 100.0 | 100.0 | 90.2
  No Worsening in PhGA | 97.4 | 97.5 | 93.1
  Treatment Failure | 0 | 2.8 | 4.9
Statistical Analysis 1: Comparison: PF-04236921 10 Milligram (10 mg) vs Placebo; >=4 points reduction in SLEDAI score: Point estimates of the ORs as well as their confidence intervals were calculated from the generalized linear mix model that included fixed factors of the stratification factors, treatment, visit and treatment by visit; Test type: Superiority; p = 0.205, Mixed Models Analysis — P-value was displayed without adjusting for multiplicity; Odds Ratio (OR) = 1.59, 90% CI 2-sided [0.63 to 4.02]
Statistical Analysis 2: Comparison: PF-04236921 50 mg vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.625, Mixed Models Analysis — P-value was displayed without adjusting for multiplicity; Odds Ratio (OR) = 0.84, 90% CI 2-sided [0.34 to 2.08]
Statistical Analysis 3: Comparison: PF-04236921 10 Milligram (10 mg) vs Placebo; No worsening in PhGA: Point estimates of the ORs as well as their confidence intervals were calculated from the generalized linear mix model that included fixed factors of the stratification factors, treatment, visit and treatment by visit; Test type: Superiority; p = 0.198, Mixed Models Analysis — P-value was displayed without adjusting for multiplicity; Odds Ratio (OR) = 2.81, 90% CI 2-sided [0.38 to 20.65]
Statistical Analysis 4: Comparison: PF-04236921 50 mg vs Placebo; [analysis description as in outcome 5, analysis 3]; Test type: Superiority; p = 0.192, Mixed Models Analysis — P-value was displayed without adjusting for multiplicity; Odds Ratio (OR) = 2.88, 90% CI 2-sided [0.39 to 21.30]

6. Secondary Outcome: Number of Participants With Clinically Significant Laboratory Tests Results
Description: Pre-defined criteria were established for each laboratory test to define the values that would be identified as of potential clinical importance. Laboratory values included Alanine Aminotransferase (ALT) [>5.0 - 10.0*Upper limit of normal range (ULN)], Albumin [<26-20 gram per liter (g/L)/ <20 g/L], Amylase [>2.0 - 5.0*ULN], Aspartate Aminotransferase (AST) [>5.0 - 10.0*ULN], Creatine Kinase (CK) [>5.0 - 10.0* ULN/ >10.0*ULN], Glucose (Hyperglycemia) [>13.9 - 27.8 millimoles/liter (mmol/L)], Hemoglobin (HGB) [<80 - 65 g/L/ <65 g/L], Lipase [>2.0 - 5.0*ULN], Lymphocytes (Lymph.)(Absolute [Abs]) [<0.5 - 0.2*10^3/microliter (UL)/ <0.2*10^3/UL], Platelets [<50-25*10^3/UL/ <25*10^3/UL], potassium (low) [<3.0 - 2.5 mmol/L], Sodium (low) [<130 - 120 mmol/L], Total Neutrophils (TN) (Abs) [<1.0 - 0.5*10^3/UL/ <0.5*10^3/UL], Triglycerides [>5.7 - 11.4 mmol/L], White Blood Cell Count (WBC) [<2.0 - 1.0*10^3/UL/ <1.0*10^3/UL].
Time Frame: Baseline up to Week 52
Population: Safety population defined as all participants who had at least one dose of investigational product. Here, "number analyzed" signifies those participants who were evaluable at specified time points.
Measure: Number; unit: Participants
Arm/Group | PF-04236921 10 Milligram (10 mg) | PF-04236921 50 mg | PF-04236921 200 mg | Placebo
Number analyzed (Participants) | 45 | 47 | 46 | 45
Participants
  ALT: number analyzed (Participants) | 45 | 47 | 45 | 45
  ALT | 2 | 0 | 0 | 0
  Albumin: <26-20 g/L: number analyzed (Participants) | 45 | 47 | 45 | 45
  Albumin: <26-20 g/L | 1 | 1 | 1 | 1
  Albumin: < 20 g/L: number analyzed (Participants) | 45 | 47 | 45 | 45
  Albumin: < 20 g/L | 0 | 1 | 0 | 0
  Amylase: number analyzed (Participants) | 45 | 47 | 45 | 45
  Amylase | 1 | 1 | 1 | 1
  AST: number analyzed (Participants) | 45 | 47 | 45 | 45
  AST | 0 | 1 | 0 | 1
  CK: >5.0 -10.0*ULN: number analyzed (Participants) | 45 | 47 | 45 | 45
  CK: >5.0 -10.0*ULN | 0 | 1 | 1 | 0
  CK >10.0*ULN: number analyzed (Participants) | 45 | 47 | 45 | 45
  CK >10.0*ULN | 0 | 1 | 1 | 0
  Glucose (Hyperglycemia): number analyzed (Participants) | 45 | 47 | 45 | 45
  Glucose (Hyperglycemia) | 1 | 1 | 0 | 2
  HGB: <80 - 65 g/L: number analyzed (Participants) | 45 | 47 | 45 | 45
  HGB: <80 - 65 g/L | 1 | 0 | 0 | 1
  HGB: <65 g/L: number analyzed (Participants) | 45 | 47 | 45 | 45
  HGB: <65 g/L | 1 | 0 | 0 | 0
  Lipase: number analyzed (Participants) | 45 | 47 | 45 | 45
  Lipase | 0 | 1 | 1 | 0
  Lymph.(Abs)<0.5-0.2* 10^3/UL: number analyzed (Participants) | 45 | 47 | 45 | 45
  Lymph.(Abs)<0.5-0.2* 10^3/UL | 6 | 9 | 4 | 8
  Lymph.(Abs) <0.2*10^3/UL: number analyzed (Participants) | 45 | 47 | 45 | 45
  Lymph.(Abs) <0.2*10^3/UL | 1 | 0 | 0 | 0
  Platelets <50 - 25*10^3/UL: number analyzed (Participants) | 45 | 47 | 45 | 45
  Platelets <50 - 25*10^3/UL | 0 | 0 | 0 | 2
  Platelets <25*10^3/UL: number analyzed (Participants) | 45 | 47 | 45 | 45
  Platelets <25*10^3/UL | 0 | 0 | 0 | 1
  Potassium (low): number analyzed (Participants) | 45 | 47 | 45 | 45
  Potassium (low) | 2 | 1 | 1 | 1
  Sodium (low): number analyzed (Participants) | 45 | 47 | 45 | 45
  Sodium (low) | 0 | 0 | 1 | 0
  TN (Abs)<1.0-0.5*10^3/UL: number analyzed (Participants) | 45 | 47 | 45 | 45
  TN (Abs)<1.0-0.5*10^3/UL | 4 | 5 | 3 | 2
  TN (Abs) <0.5*10^3/UL: number analyzed (Participants) | 45 | 47 | 45 | 45
  TN (Abs) <0.5*10^3/UL | 1 | 1 | 1 | 0
  Triglycerides: number analyzed (Participants) | 44 | 47 | 45 | 45
  Triglycerides | 0 | 1 | 0 | 2
  WBC <2.0 - 1.0*10^3/UL: number analyzed (Participants) | 45 | 47 | 45 | 45
  WBC <2.0 - 1.0*10^3/UL | 4 | 2 | 2 | 2
  WBC <1.0*10^3/UL: number analyzed (Participants) | 45 | 47 | 45 | 45
  WBC <1.0*10^3/UL | 1 | 0 | 0 | 0

7. Secondary Outcome: Number of Participants Who Discontinued Due to Adverse Events
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Number of participants who discontinued due to adverse events were reported.
Time Frame: Baseline up to Week 52
Population: Safety population defined as all participants who had at least one dose of investigational product.
Measure: Number; unit: Participants
Arm/Group | PF-04236921 10 Milligram (10 mg) | PF-04236921 50 mg | PF-04236921 200 mg | Placebo
Number analyzed (Participants) | 45 | 47 | 46 | 45
Participants | 3 | 2 | 3 | 3

8. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) or Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to Week 52 that were absent before treatment or that worsened relative to pretreatment state. Number of participants with treatment-emergent AEs or SAEs (excluding infectious AEs or SAEs and injection site reactions) were reported. AEs include both SAEs and non-SAEs.
Time Frame: Baseline up to Week 52
Population: Safety population defined as all participants who had at least one dose of investigational product.
Measure: Number; unit: Participants
Arm/Group | PF-04236921 10 Milligram (10 mg) | PF-04236921 50 mg | PF-04236921 200 mg | Placebo
Number analyzed (Participants) | 45 | 47 | 46 | 45
Participants
  AEs | 34 | 36 | 38 | 40
  SAEs | 4 | 2 | 7 | 8

9. Secondary Outcome: Number of Participants With Treatment-Emergent Infectious Adverse Events (AEs) or Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to Week 52 that were absent before treatment or that worsened relative to pretreatment state. Number of participants with treatment-emergent infectious AEs or SAEs were reported. AEs include both SAEs and non-SAEs.
Time Frame: Baseline up to Week 52
Population: Safety population defined as all participants who had at least one dose of investigational product.
Measure: Number; unit: Participants
Arm/Group | PF-04236921 10 Milligram (10 mg) | PF-04236921 50 mg | PF-04236921 200 mg | Placebo
Number analyzed (Participants) | 45 | 47 | 46 | 45
Participants
  Infectious AEs | 25 | 28 | 25 | 26
  Infectious SAEs | 2 | 3 | 4 | 4

10. Secondary Outcome: Number of Participants With Potentially Clinically Important (PCI) Electrocardiogram (ECG) Findings
Description: Criteria for potentially clinically important (PCI) findings in ECG were defined as: heart rate <=40 beats per minute (bpm) or >=120 bpm; PR interval >=220 millisecond (msec); QT interval >=480 msec; QRS interval >=120 msec; QT interval corrected using the Fridericia formula (QTcF) >=500msec; no sinus rhythm.
Time Frame: Baseline up to Week 52
Population: Safety population defined as all participants who had at least one dose of investigational product. Here, N (Number of participants analyzed) signifies participants evaluable for this outcome measure for each group respectively.
Measure: Number; unit: Participants
Arm/Group | PF-04236921 10 Milligram (10 mg) | PF-04236921 50 mg | PF-04236921 200 mg | Placebo
Number analyzed (Participants) | 42 | 46 | 44 | 44
Participants
  Heart Rate <=40 beats/min or >=120 beats/min | 0 | 0 | 0 | 0
  PR Interval >=200 msec | 2 | 1 | 1 | 2
  QT Interval >=480 msec | 2 | 0 | 0 | 0
  QRS Interval >=120 msec | 3 | 1 | 2 | 2
  QTcF >=500 msec | 2 | 0 | 0 | 0
  Rhythm (Not Sinus Rhythm) | 0 | 0 | 0 | 1

11. Secondary Outcome: Number of Participants With Potentially Clinically Important Vital Signs Findings
Description: Criteria for PCI findings in vital signs were defined as: sitting systolic blood pressure (Increase from baseline >=20 millimeter of mercury (mm Hg) and >=160 mm Hg or a decrease from baseline >=20 mm Hg and <=90 mm Hg) and sitting diastolic blood pressure (increase from baseline >=15 mm Hg and >=90 mm Hg or decrease from baseline >=15 mm Hg and <=60 mm Hg), pulse rate (increase from baseline >=15 beats/min and >=120 beats/min or decrease from baseline >=15 beats/min and <=50 beats /min), body temperature (increase of >=2 degree Fahrenheit (F) and temperature >=101 degree F) and weight (change of >=7% in body weight)
Time Frame: Baseline up to Week 52
Population: Safety population defined as all participants who had at least one dose of investigational product.
Measure: Number; unit: Participants
Arm/Group | PF-04236921 10 Milligram (10 mg) | PF-04236921 50 mg | PF-04236921 200 mg | Placebo
Number analyzed (Participants) | 45 | 47 | 46 | 45
Participants
  Sitting Systolic Blood Pressure | 8 | 3 | 3 | 5
  Sitting Diastolic Blood Pressure | 14 | 14 | 12 | 14
  Sitting Pulse Rate | 1 | 1 | 0 | 1
  Temperature | 0 | 0 | 0 | 0
  Weight | 12 | 23 | 14 | 14

12. Secondary Outcome: Number of Participants With Anti-drug Antibodies (ADAs) and Neutralizing Antibodies (Nabs)
Description: Human serum samples were analyzed for the presence or absence of anti-PF-04236921 antibodies. A positive ADA sample was further tested for neutralizing antibodies using a validated assay.
Time Frame: Baseline up to Week 52
Population: Safety population defined as all participants who had at least one dose of investigational product.
Measure: Number; unit: Participants
Arm/Group | PF-04236921 10 Milligram (10 mg) | PF-04236921 50 mg | PF-04236921 200 mg | Placebo
Number analyzed (Participants) | 45 | 47 | 46 | 45
Participants
  Anti-drug Antibodies | 1 | 0 | 1 | 0
  Neutralizing Antibodies | 0 | 0 | 0 | 0

13. Secondary Outcome: Serum Concentration of PF-04236921
Description: Serum PF-04236921 concentrations over time were summarized.
Time Frame: Day 1, Week 2, 4, 6, 8, 12, 16, 20, 24
Population: Pharmacokinetic analysis set was the subset of participants from safety analysis set (all participants who received at least 1 dose of investigational product) who provided at least 1 pharmacokinetic concentration. Here, "number analyzed" signifies those participants who were evaluable at specified time points.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | PF-04236921 10 Milligram (10 mg) | PF-04236921 50 mg | PF-04236921 200 mg
Number analyzed (Participants) | 45 | 47 | 46
nanogram per milliliter (ng/mL)
  Day 1: number analyzed (Participants) | 42 | 45 | 43
  Day 1 | 26.3 (110.8) | 31.0 (146.9) | 15.2 (99.8)
  Week 2: number analyzed (Participants) | 37 | 41 | 40
  Week 2 | 1297 (759.4) | 5640 (2274.0) | 22780 (9896.0)
  Week 4: number analyzed (Participants) | 39 | 42 | 38
  Week 4 | 991.8 (527.6) | 4337 (1495.0) | 17550 (5757.1)
  Week 6: number analyzed (Participants) | 39 | 40 | 37
  Week 6 | 608.4 (330.1) | 3396 (1410.0) | 13460 (5416.6)
  Week 8: number analyzed (Participants) | 39 | 38 | 30
  Week 8 | 463.4 (254.9) | 2709 (1317.5) | 11110 (5023.7)
  Week 12: number analyzed (Participants) | 32 | 33 | 28
  Week 12 | 1210 (607.0) | 6482 (2487.4) | 25240 (8114.0)
  Week 16: number analyzed (Participants) | 31 | 36 | 23
  Week 16 | 703.2 (407.4) | 3886 (1322.1) | 16990 (6203.4)
  Week 20: number analyzed (Participants) | 30 | 34 | 17
  Week 20 | 1452 (726.8) | 6978 (2954.0) | 31050 (11368)
  Week 24: number analyzed (Participants) | 31 | 34 | 18
  Week 24 | 871.9 (450.4) | 4417 (2402.4) | 20150 (12091)

14. Secondary Outcome: Percentage of Participants With Corticosteroid Dose Reduced by Both Greater Than or Equal to (>=) 25 Percent (%) From Baseline and Less Than or Equal to (<=) 7.5 Milligrams Per Day (mg/Day)
Description: Participants were given supplemental corticosteroids at baseline to control disease activity, if necessary. The steroid taper was based on participant's symptoms. Participants recorded their steroid usage on a diary card. Least Observation Carried Forward (LOCF) method was used to impute missing data.
Time Frame: Week 12, 16, 20, 24
Population: Full Analysis Set= all randomized participants who received at least 1 dose of study drug. Number of participants analyzed= participants evaluable for this outcome measure at specified timepoints. As per sponsor's decision, dosing in "PF-04236921 200 mg" arm was prematurely terminated and hence it was not included in efficacy analysis.
Measure: Number; unit: Percentage of Participants
Arm/Group | PF-04236921 10 Milligram (10 mg) | PF-04236921 50 mg | Placebo
Number analyzed (Participants) | 15 | 24 | 23
Percentage of Participants
  Week 12 | 13.3 | 20.8 | 8.7
  Week 16 | 20.0 | 25.0 | 8.7
  Week 20 | 26.7 | 25.0 | 8.7
  Week 24 | 26.7 | 20.8 | 8.7

15. Secondary Outcome: Percentage of Participants With Normalized Serological Activity
Description: Serologic activity was to be assessed in the subgroup of participants who had positive serologic activity at baseline.
Time Frame: Baseline up to Week 24
Population: Consistent with the protocol which pre-specified that if the number of participants with abnormal serological activity at baseline were <25% of overall population, data for this outcome measure was not available.
Arm/Group | PF-04236921 10 Milligram (10 mg) | PF-04236921 50 mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0

16. Secondary Outcome: Patient Global Visual Analog Scale (VAS) Scores at Baseline
Description: Participants assessed their disease activity using a 100 millimeter (mm) VAS. Participants answered the following question "Considering all the ways your disease affects you, how are you feeling today?" Response was recorded by placing a mark on the scale between 0 (very well) and 100 (extremely bad).
Time Frame: Baseline
Population: Full Analysis Set= all randomized participants who received at least 1 dose of study drug. As per sponsor's decision, dosing in "PF-04236921 200 mg" arm was prematurely terminated and hence it was not included in efficacy analysis.
Measure: Mean (Standard Error); unit: mm
Arm/Group | PF-04236921 10 Milligram (10 mg) | PF-04236921 50 mg | Placebo
Number analyzed (Participants) | 45 | 47 | 45
mm | 50.44 (2.865) | 47.70 (2.880) | 49.47 (3.349)

17. Secondary Outcome: Change From Baseline in Patient Global Visual Analog Scale (VAS) at Week 2, 4, 6, 8, 12, 16, 20 and 24
Description: Participants assessed their disease activity using a 100 mm VAS. Participants answered the following question "Considering all the ways your disease affects you, how are you feeling today?" Response was recorded by placing a mark on the scale between 0 (very well) and 100 (extremely bad).
Time Frame: Baseline, Week 2, 4, 6, 8, 12, 16, 20, 24
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: mm
Arm/Group | PF-04236921 10 Milligram (10 mg) | PF-04236921 50 mg | Placebo
Number analyzed (Participants) | 45 | 47 | 45
mm
  Week 2: number analyzed (Participants) | 44 | 47 | 43
  Week 2 | -9.17 [-15.09 to -3.26] | -1.54 [-7.22 to 4.15] | -3.58 [-9.49 to 2.34]
  Week 4 | -3.24 [-9.09 to 2.62] | -4.01 [-9.69 to 1.68] | -1.24 [-7.02 to 4.55]
  Week 6 | -5.48 [-11.33 to 0.37] | -3.62 [-9.31 to 2.06] | -7.24 [-13.02 to -1.45]
  Week 8 | -4.17 [-10.02 to 1.68] | -6.03 [-11.71 to -0.34] | -7.11 [-12.89 to -1.32]
  Week 12 | -9.21 [-15.07 to -3.36] | -4.20 [-9.88 to 1.49] | -6.88 [-12.67 to -1.10]
  Week 16 | -8.75 [-14.60 to -2.89] | -10.20 [-15.88 to -4.51] | -5.99 [-11.78 to -0.21]
  Week 20 | -11.52 [-17.38 to -5.67] | -9.03 [-14.71 to -3.34] | -6.77 [-12.56 to -0.99]
  Week 24 | -9.17 [-15.02 to -3.32] | -7.45 [-13.14 to -1.77] | -10.64 [-16.42 to -4.85]
Statistical Analysis 1: Comparison: PF-04236921 10 Milligram (10 mg) vs Placebo; Week 2: Analysis was done using linear mixed effect model that included fixed factors of the stratification factors, treatment, visit, treatment by visit and baseline VAS; Test type: Superiority; LS mean difference = -5.41, 90% CI 2-sided [-12.30 to 1.49]
Statistical Analysis 2: Comparison: PF-04236921 10 Milligram (10 mg) vs Placebo; Week 4: Analysis was done using linear mixed effect model that included fixed factors of the stratification factors, treatment, visit, treatment by visit and baseline VAS; Test type: Superiority; LS Mean difference = -1.39, 90% CI 2-sided [-8.21 to 5.42]
Statistical Analysis 3: Comparison: PF-04236921 10 Milligram (10 mg) vs Placebo; Week 6: Analysis was done using linear mixed effect model that included fixed factors of the stratification factors, treatment, visit, treatment by visit and baseline VAS; Test type: Superiority; LS Mean difference = 1.30, 90% CI 2-sided [-5.71 to 8.32]
Statistical Analysis 4: Comparison: PF-04236921 10 Milligram (10 mg) vs Placebo; Week 8: Analysis was done using linear mixed effect model that included fixed factors of the stratification factors, treatment, visit, treatment by visit and baseline VAS; Test type: Superiority; LS Mean difference = 4.67, 90% CI 2-sided [-2.22 to 11.57]
Statistical Analysis 5: Comparison: PF-04236921 10 Milligram (10 mg) vs Placebo; Week 12: Analysis was done using linear mixed effect model that included fixed factors of the stratification factors, treatment, visit, treatment by visit and baseline VAS; Test type: Superiority; LS Mean difference = -3.98, 90% CI 2-sided [-11.04 to 3.07]
Statistical Analysis 6: Comparison: PF-04236921 10 Milligram (10 mg) vs Placebo; Week 16: Analysis was done using linear mixed effect model that included fixed factors of the stratification factors, treatment, visit, treatment by visit and baseline VAS; Test type: Superiority; LS Mean difference = -2.89, 90% CI 2-sided [-9.87 to 4.10]
Statistical Analysis 7: Comparison: PF-04236921 10 Milligram (10 mg) vs Placebo; Week 20: Analysis was done using linear mixed effect model that included fixed factors of the stratification factors, treatment, visit, treatment by visit and baseline VAS; Test type: Superiority; LS Mean difference = -6.21, 90% CI 2-sided [-13.37 to 0.94]
Statistical Analysis 8: Comparison: PF-04236921 10 Milligram (10 mg) vs Placebo; Week 24: Analysis was done using linear mixed effect model that included fixed factors of the stratification factors, treatment, visit, treatment by visit and baseline VAS; Test type: Superiority; LS Mean difference = 1.98, 90% CI 2-sided [-5.17 to 9.13]
Statistical Analysis 9: Comparison: PF-04236921 50 mg vs Placebo; [analysis description as in outcome 17, analysis 1]; Test type: Superiority; LS Mean difference = 2.07, 90% CI 2-sided [-4.70 to 8.84]
Statistical Analysis 10: Comparison: PF-04236921 50 mg vs Placebo; [analysis description as in outcome 17, analysis 2]; Test type: Superiority; LS Mean difference = -2.81, 90% CI 2-sided [-9.62 to 4.00]
Statistical Analysis 11: Comparison: PF-04236921 50 mg vs Placebo; [analysis description as in outcome 17, analysis 3]; Test type: Superiority; LS Mean difference = 3.97, 90% CI 2-sided [-2.95 to 10.90]
Statistical Analysis 12: Comparison: PF-04236921 50 mg vs Placebo; [analysis description as in outcome 17, analysis 4]; Test type: Superiority; LS Mean difference = 2.56, 90% CI 2-sided [-4.29 to 9.40]
Statistical Analysis 13: Comparison: PF-04236921 50 mg vs Placebo; [analysis description as in outcome 17, analysis 5]; Test type: Superiority; LS Mean difference = 3.14, 90% CI 2-sided [-3.67 to 9.94]
Statistical Analysis 14: Comparison: PF-04236921 50 mg vs Placebo; [analysis description as in outcome 17, analysis 6]; Test type: Superiority; LS Mean difference = -4.94, 90% CI 2-sided [-11.91 to 2.03]
Statistical Analysis 15: Comparison: PF-04236921 50 mg vs Placebo; [analysis description as in outcome 17, analysis 7]; Test type: Superiority; LS Mean difference = -2.64, 90% CI 2-sided [-9.61 to 4.32]
Statistical Analysis 16: Comparison: PF-04236921 50 mg vs Placebo; [analysis description as in outcome 17, analysis 8]; Test type: Superiority; LS Mean difference = 2.66, 90% CI 2-sided [-4.48 to 9.80]

18. Secondary Outcome: Change From Baseline in European Quality of Life 5 Dimensions Questionnaire (EQ-5D) at Week 4, 8, 12, 16, 20 and 24
Description: EQ-5D is a standardized, participant-administered measure of health outcome. It provides a descriptive profile for 5 dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression), using 3 levels (no, moderate, or extreme problems) and a single index value characterizing current health status using a 100-point VAS (0= worst imaginable health state, 100= best imaginable health state).
Time Frame: Baseline, Week 4, 8, 12, 16, 20, 24
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | PF-04236921 10 Milligram (10 mg) | PF-04236921 50 mg | Placebo
Number analyzed (Participants) | 45 | 47 | 45
Units on a scale
  Week 4: number analyzed (Participants) | 43 | 46 | 45
  Week 4 | 3.17 [-2.21 to 8.54] | 1.45 [-3.72 to 6.62] | -0.47 [-5.66 to 4.73]
  Week 8: number analyzed (Participants) | 43 | 47 | 45
  Week 8 | 5.00 [-0.37 to 10.38] | 2.82 [-2.28 to 7.93] | 7.02 [1.83 to 12.22]
  Week 12: number analyzed (Participants) | 43 | 47 | 45
  Week 12 | 7.47 [2.09 to 12.85] | 2.51 [-2.60 to 7.61] | 4.85 [-0.35 to 10.04]
  Week 16: number analyzed (Participants) | 43 | 47 | 45
  Week 16 | 6.84 [1.47 to 12.22] | 6.65 [1.55 to 11.76] | 5.16 [-0.04 to 10.35]
  Week 20: number analyzed (Participants) | 43 | 47 | 45
  Week 20 | 9.68 [4.30 to 15.05] | 5.19 [0.08 to 10.29] | 5.09 [-0.10 to 10.28]
  Week 24: number analyzed (Participants) | 43 | 47 | 45
  Week 24 | 9.33 [3.95 to 14.71] | 5.04 [-0.07 to 10.14] | 5.38 [0.18 to 10.57]
Statistical Analysis 1: Comparison: PF-04236921 10 Milligram (10 mg) vs Placebo; Week 4: Analysis was done using linear mixed effect model that included fixed factors of the stratification factors, treatment, visit, treatment by visit and baseline tender score; Test type: Superiority; LS mean difference = 3.63, 90% CI [-2.56 to 9.83]
Statistical Analysis 2: Comparison: PF-04236921 10 Milligram (10 mg) vs Placebo; Week 8: Analysis was done using linear mixed effect model that included fixed factors of the stratification factors, treatment, visit, treatment by visit and baseline tender score; Test type: Superiority; LS mean difference = -2.02, 90% CI [-8.21 to 4.18]
Statistical Analysis 3: Comparison: PF-04236921 10 Milligram (10 mg) vs Placebo; Week 12: Analysis was done using linear mixed effect model that included fixed factors of the stratification factors, treatment, visit, treatment by visit and baseline tender score; Test type: Superiority; LS mean difference = 2.62, 90% CI 2-sided [-3.57 to 8.82]
Statistical Analysis 4: Comparison: PF-04236921 10 Milligram (10 mg) vs Placebo; Week 16: Analysis was done using linear mixed effect model that included fixed factors of the stratification factors, treatment, visit, treatment by visit and baseline tender score; Test type: Superiority; LS mean difference = 1.69, 90% CI 2-sided [-4.51 to 7.88]
Statistical Analysis 5: Comparison: PF-04236921 10 Milligram (10 mg) vs Placebo; Week 20: Analysis was done using linear mixed effect model that included fixed factors of the stratification factors, treatment, visit, treatment by visit and baseline tender score; Test type: Superiority; LS mean difference = 4.59, 90% CI 2-sided [-1.61 to 10.79]
Statistical Analysis 6: Comparison: PF-04236921 10 Milligram (10 mg) vs Placebo; Week 24: Analysis was done using linear mixed effect model that included fixed factors of the stratification factors, treatment, visit, treatment by visit and baseline tender score; Test type: Superiority; LS mean difference = 3.95, 90% CI [-2.24 to 10.15]
Statistical Analysis 7: Comparison: PF-04236921 50 mg vs Placebo; [analysis description as in outcome 18, analysis 1]; Test type: Superiority; LS mean difference = 1.92, 90% CI [-4.17 to 8.01]
Statistical Analysis 8: Comparison: PF-04236921 50 mg vs Placebo; [analysis description as in outcome 18, analysis 2]; Test type: Superiority; LS mean difference = -4.20, 90% CI [-10.25 to 1.85]
Statistical Analysis 9: Comparison: PF-04236921 50 mg vs Placebo; [analysis description as in outcome 18, analysis 4]; Test type: Superiority; LS mean difference = 1.50, 90% CI 2-sided [-4.56 to 7.55]
Statistical Analysis 10: Comparison: PF-04236921 50 mg vs Placebo; [analysis description as in outcome 18, analysis 5]; Test type: Superiority; LS mean difference = 0.10, 90% CI 2-sided [-5.96 to 6.15]
Statistical Analysis 11: Comparison: PF-04236921 50 mg vs Placebo; [analysis description as in outcome 18, analysis 6]; Test type: Superiority; LS mean difference = -0.34, 90% CI 2-sided [-6.39 to 5.71]
Statistical Analysis 12: Comparison: PF-04236921 50 mg vs Placebo; [analysis description as in outcome 18, analysis 3]; Test type: Superiority; LS mean difference = -2.34, 90% CI 2-sided [-8.39 to 3.71]

19. Secondary Outcome: Thirty Six-Item Short-Form Health Survey (SF-36) Physical Component Score (PCS) and Mental Component Score (MCS) at Baseline
Description: SF-36 is a standardized survey evaluating 8 aspects of functional health and well-being: physical and social functioning, physical and emotional role limitations, bodily pain, general health, vitality, mental health. These 8 aspects can also be summarized as PCS and mental component score MCS. The score for each aspect and PCS/MCS is an average of the individual question scores, which are scaled 0-100 (100=highest level of functioning). LOCF method was used to impute missing values.
Time Frame: Baseline
Population: Full Analysis Set= all randomized participants who received at least 1 dose of study drug. Number of participants analyzed= participants evaluable for this outcome measure at specified timepoint. As per sponsor's decision, dosing in "PF-04236921 200 mg" arm was prematurely terminated and hence it was not included in efficacy analysis.
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | PF-04236921 10 Milligram (10 mg) | PF-04236921 50 mg | Placebo
Number analyzed (Participants) | 43 | 46 | 45
Units on a scale
  MCS | 39.50 (1.810) | 42.36 (1.426) | 39.94 (1.450)
  PCS | 33.47 (1.169) | 34.36 (1.250) | 34.64 (1.523)

20. Secondary Outcome: Change From Baseline in 36-Item Short-Form Health Survey (SF-36) PCS and MCS at Week 4, 8, 12, 16, 20 and 24
Description: SF-36 is a standardized survey evaluating 8 aspects of functional health and well-being: physical and social functioning, physical and emotional role limitations, bodily pain, general health, vitality, mental health. These 8 aspects can also be summarized as physical component score (PCS) and mental component score (MCS). The score for each aspect and PCS/MCS is an average of the individual question scores, which are scaled 0-100 (100=highest level of functioning). LOCF method was used to impute missing values.
Time Frame: Baseline, Week 4, 8, 12, 16, 20, 24
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | PF-04236921 10 Milligram (10 mg) | PF-04236921 50 mg | Placebo
Number analyzed (Participants) | 45 | 47 | 45
Units on a scale
  MCS: Week 4: number analyzed (Participants) | 43 | 45 | 45
  MCS: Week 4 | 1.97 [-0.69 to 4.64] | 1.45 [-1.14 to 4.04] | 1.45 [-1.12 to 4.02]
  MCS: Week 8: number analyzed (Participants) | 43 | 46 | 45
  MCS: Week 8 | 1.57 [-1.10 to 4.23] | 1.97 [-0.59 to 4.52] | 2.05 [-0.52 to 4.62]
  MCS: Week 12: number analyzed (Participants) | 43 | 46 | 45
  MCS: Week 12 | 3.80 [1.13 to 6.46] | 2.50 [-0.06 to 5.05] | 2.52 [-0.05 to 5.09]
  MCS: Week 16: number analyzed (Participants) | 43 | 46 | 45
  MCS: Week 16 | 4.73 [2.07 to 7.40] | 2.79 [0.24 to 5.35] | 2.95 [0.38 to 5.52]
  MCS: Week 20: number analyzed (Participants) | 43 | 46 | 45
  MCS: Week 20 | 4.49 [1.82 to 7.15] | 1.71 [-0.85 to 4.26] | 3.28 [0.71 to 5.85]
  MCS: Week 24: number analyzed (Participants) | 43 | 46 | 45
  MCS: Week 24 | 2.94 [0.28 to 5.60] | 2.14 [-0.41 to 4.70] | 2.85 [0.28 to 5.42]
  PCS: Week 4: number analyzed (Participants) | 43 | 45 | 45
  PCS: Week 4 | 3.95 [1.75 to 6.15] | 3.24 [1.10 to 5.38] | 1.28 [-0.85 to 3.40]
  PCS: Week 8: number analyzed (Participants) | 43 | 46 | 45
  PCS: Week 8 | 5.48 [3.27 to 7.68] | 4.79 [2.68 to 6.90] | 2.11 [-0.01 to 4.23]
  PCS: Week 12: number analyzed (Participants) | 43 | 46 | 45
  PCS: Week 12 | 6.06 [3.86 to 8.26] | 4.66 [2.55 to 6.77] | 2.82 [0.70 to 4.95]
  PCS: Week 16: number analyzed (Participants) | 43 | 46 | 45
  PCS: Week 16 | 6.25 [4.05 to 8.45] | 4.50 [2.39 to 6.61] | 2.48 [0.36 to 4.60]
  PCS: Week 20: number analyzed (Participants) | 43 | 46 | 45
  PCS: Week 20 | 6.39 [4.19 to 8.59] | 5.63 [3.52 to 7.74] | 3.29 [1.17 to 5.42]
  PCS: Week 24: number analyzed (Participants) | 43 | 46 | 45
  PCS: Week 24 | 5.98 [3.77 to 8.18] | 5.53 [3.42 to 7.64] | 2.94 [0.82 to 5.06]
Statistical Analysis 1: Comparison: PF-04236921 10 Milligram (10 mg) vs Placebo; MCS Week 4: Analysis was done using the ANCOVA model; CI parameter being the LS mean difference from that model; Test type: Superiority; LS mean difference = 0.53, 90% CI 2-sided [-2.53 to 3.59]
Statistical Analysis 2: Comparison: PF-04236921 10 Milligram (10 mg) vs Placebo; MCS Week 8: Analysis was done using the ANCOVA model; CI parameter being the LS mean difference from that model; Test type: Superiority; LS mean difference = -0.48, 90% CI 2-sided [-3.54 to 2.58]
Statistical Analysis 3: Comparison: PF-04236921 10 Milligram (10 mg) vs Placebo; MCS Week 12: Analysis was done using the ANCOVA model; CI parameter being the LS mean difference from that model; Test type: Superiority; LS mean difference = 1.28, 90% CI 2-sided [-1.78 to 4.34]
Statistical Analysis 4: Comparison: PF-04236921 10 Milligram (10 mg) vs Placebo; MCS Week 16: Analysis was done using the ANCOVA model; CI parameter being the LS mean difference from that model; Test type: Superiority; LS mean difference = 1.78, 90% CI 2-sided [-1.28 to 4.84]
Statistical Analysis 5: Comparison: PF-04236921 10 Milligram (10 mg) vs Placebo; MCS Week 20: Analysis was done using the ANCOVA model; CI parameter being the LS mean difference from that model; Test type: Superiority; LS mean difference = 1.20, 90% CI 2-sided [-1.86 to 4.26]
Statistical Analysis 6: Comparison: PF-04236921 10 Milligram (10 mg) vs Placebo; MCS Week 24: Analysis was done using the ANCOVA model; CI parameter being the LS mean difference from that model; Test type: Superiority; LS mean difference = 0.09, 90% CI 2-sided [-2.98 to 3.15]
Statistical Analysis 7: Comparison: PF-04236921 50 mg vs Placebo; MCS Week 4: Analysis was done using the ANCOVA model; CI parameter being the LS mean difference from that model; Test type: Superiority; LS mean difference = 0.00, 90% CI 2-sided [-3.03 to 3.03]
Statistical Analysis 8: Comparison: PF-04236921 50 mg vs Placebo; MCS Week 8: Analysis was done using the ANCOVA model; CI parameter being the LS mean difference from that model; Test type: Superiority; LS mean difference = -0.09, 90% CI 2-sided [-3.09 to 2.92]
Statistical Analysis 9: Comparison: PF-04236921 50 mg vs Placebo; MCS Week 12: Analysis was done using the ANCOVA model; CI parameter being the LS mean difference from that model; Test type: Superiority; LS mean difference = -0.02, 90% CI 2-sided [-3.03 to 2.99]
Statistical Analysis 10: Comparison: PF-04236921 50 mg vs Placebo; MCS Week 16: Analysis was done using the ANCOVA model; CI parameter being the LS mean difference from that model; Test type: Superiority; LS mean difference = -0.16, 90% CI 2-sided [-3.17 to 2.85]
Statistical Analysis 11: Comparison: PF-04236921 50 mg vs Placebo; MCS Week 20: Analysis was done using the ANCOVA model; CI parameter being the LS mean difference from that model; Test type: Superiority; LS mean difference = -1.58, 90% CI 2-sided [-4.58 to 1.43]
Statistical Analysis 12: Comparison: PF-04236921 50 mg vs Placebo; MCS Week 24: Analysis was done using the ANCOVA model; CI parameter being the LS mean difference from that model; Test type: Superiority; LS mean difference = -0.71, 90% CI 2-sided [-3.72 to 2.30]
Statistical Analysis 13: Comparison: PF-04236921 10 Milligram (10 mg) vs Placebo; PCS Week 4: Analysis was done using the ANCOVA model; CI parameter being the LS mean difference from that model; Test type: Superiority; LS mean difference = 2.67, 90% CI 2-sided [0.14 to 5.20]
Statistical Analysis 14: Comparison: PF-04236921 10 Milligram (10 mg) vs Placebo; PCS Week 8: Analysis was done using the ANCOVA model; CI parameter being the LS mean difference from that model; Test type: Superiority; LS mean difference = 3.36, 90% CI 2-sided [0.84 to 5.89]
Statistical Analysis 15: Comparison: PF-04236921 10 Milligram (10 mg) vs Placebo; PCS Week 12: Analysis was done using the ANCOVA model; CI parameter being the LS mean difference from that model; Test type: Superiority; LS mean difference = 3.23, 90% CI 2-sided [0.70 to 5.76]
Statistical Analysis 16: Comparison: PF-04236921 10 Milligram (10 mg) vs Placebo; PCS Week 16: Analysis was done using the ANCOVA model; CI parameter being the LS mean difference from that model; Test type: Superiority; LS mean difference = 3.77, 90% CI 2-sided [1.24 to 6.30]
Statistical Analysis 17: Comparison: PF-04236921 10 Milligram (10 mg) vs Placebo; PCS Week 20: Analysis was done using the ANCOVA model; CI parameter being the LS mean difference from that model; Test type: Superiority; LS mean difference = 3.10, 90% CI 2-sided [0.57 to 5.63]
Statistical Analysis 18: Comparison: PF-04236921 10 Milligram (10 mg) vs Placebo; PCS Week 24: Analysis was done using the ANCOVA model; CI parameter being the LS mean difference from that model; Test type: Superiority; LS mean difference = 3.03, 90% CI [0.50 to 5.56]
Statistical Analysis 19: Comparison: PF-04236921 50 mg vs Placebo; PCS Week 4: Analysis was done using the ANCOVA model; CI parameter being the LS mean difference from that model; Test type: Superiority; LS mean difference = 1.96, 90% CI 2-sided [-0.53 to 4.46]
Statistical Analysis 20: Comparison: PF-04236921 50 mg vs Placebo; PCS Week 8: Analysis was done using the ANCOVA model; CI parameter being the LS mean difference from that model; Test type: Superiority; LS mean difference = 2.68, 90% CI [0.20 to 5.17]
Statistical Analysis 21: Comparison: PF-04236921 50 mg vs Placebo; PCS Week 12: Analysis was done using the ANCOVA model; CI parameter being the LS mean difference from that model; Test type: Superiority; LS mean difference = 1.84, 90% CI 2-sided [-0.65 to 4.32]
Statistical Analysis 22: Comparison: PF-04236921 50 mg vs Placebo; PCS Week 16: Analysis was done using the ANCOVA model; CI parameter being the LS mean difference from that model; Test type: Superiority; LS mean difference = 2.01, 90% CI 2-sided [-0.47 to 4.50]
Statistical Analysis 23: Comparison: PF-04236921 50 mg vs Placebo; PCS Week 20: Analysis was done using the ANCOVA model; CI parameter being the LS mean difference from that model; Test type: Superiority; LS mean difference = 2.34, 90% CI 2-sided [-0.15 to 4.82]
Statistical Analysis 24: Comparison: PF-04236921 50 mg vs Placebo; PCS Week 24: Analysis was done using the ANCOVA model; CI parameter being the LS mean difference from that model; Test type: Superiority; LS mean difference = 2.59, 90% CI 2-sided [0.11 to 5.08]

21. Secondary Outcome: Change From Baseline in Vitality Scores at Week 4, 8, 12, 16, 20 and 24
Description: SF-36 is a standardized survey evaluating 8 aspects of functional health and well being: physical and social functioning, physical and emotional role limitations, bodily pain, general health, vitality, mental health. Vitality sub-score is a component of SF-36 Health Survey Questionnaire and assesses energy and fatigue. The vitality score ranged from 0-100 (100=highest level of functioning). LOCF method was used to impute missing values.
Time Frame: Baseline, Week 4, 8, 12, 16, 20, 24
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | PF-04236921 10 Milligram (10 mg) | PF-04236921 50 mg | Placebo
Number analyzed (Participants) | 45 | 47 | 45
Units on a scale
  Week 4: number analyzed (Participants) | 43 | 45 | 45
  Week 4 | 3.92 [-2.00 to 9.83] | 4.78 [-0.97 to 10.52] | 3.45 [-2.27 to 9.16]
  Week 8: number analyzed (Participants) | 43 | 46 | 45
  Week 8 | 6.53 [0.62 to 12.45] | 6.55 [0.87 to 12.23] | 2.61 [-3.10 to 8.33]
  Week 12: number analyzed (Participants) | 43 | 46 | 45
  Week 12 | 10.75 [4.83 to 16.66] | 6.41 [0.74 to 12.09] | 7.19 [1.48 to 12.91]
  Week 16: number analyzed (Participants) | 43 | 46 | 45
  Week 16 | 10.60 [4.69 to 16.52] | 6.41 [0.74 to 12.09] | 2.75 [-2.97 to 8.46]
  Week 20: number analyzed (Participants) | 43 | 46 | 45
  Week 20 | 11.91 [5.99 to 17.82] | 7.78 [2.10 to 13.45] | 4.79 [-0.93 to 10.50]
  Week 24: number analyzed (Participants) | 43 | 46 | 45
  Week 24 | 9.58 [3.66 to 15.49] | 6.69 [1.01 to 12.37] | 5.25 [-0.47 to 10.96]
Statistical Analysis 1: Comparison: PF-04236921 10 Milligram (10 mg) vs Placebo; Week 4: Analysis was done using the ANCOVA model; CI parameter being the LS mean difference from that model; Test type: Superiority; LS mean difference = 0.47, 90% CI [-6.33 to 7.27]
Statistical Analysis 2: Comparison: PF-04236921 10 Milligram (10 mg) vs Placebo; Week 8: Analysis was done using the ANCOVA model; CI parameter being the LS mean difference from that model; Test type: Superiority; LS mean difference = 3.92, 90% CI [-2.88 to 10.72]
Statistical Analysis 3: Comparison: PF-04236921 10 Milligram (10 mg) vs Placebo; Week 12: Analysis was done using the ANCOVA model; CI parameter being the LS mean difference from that model; Test type: Superiority; LS mean difference = 3.55, 90% CI 2-sided [-3.25 to 10.36]
Statistical Analysis 4: Comparison: PF-04236921 10 Milligram (10 mg) vs Placebo; Week 16: Analysis was done using the ANCOVA model; CI parameter being the LS mean difference from that model; Test type: Superiority; LS mean difference = 7.85, 90% CI 2-sided [1.05 to 14.66]
Statistical Analysis 5: Comparison: PF-04236921 10 Milligram (10 mg) vs Placebo; Week 20: Analysis was done using the ANCOVA model; CI parameter being the LS mean difference from that model; Test type: Superiority; LS mean difference = 7.12, 90% CI 2-sided [0.32 to 13.92]
Statistical Analysis 6: Comparison: PF-04236921 10 Milligram (10 mg) vs Placebo; Week 24: Analysis was done using the ANCOVA model; CI parameter being the LS mean difference from that model; Test type: Superiority; LS mean difference = 4.33, 90% CI 2-sided [-2.47 to 11.13]
Statistical Analysis 7: Comparison: PF-04236921 50 mg vs Placebo; Week 4: Analysis was done using the ANCOVA model; CI parameter being the LS mean difference from that model; Test type: Superiority; LS mean difference = 1.33, 90% CI 2-sided [-5.40 to 8.05]
Statistical Analysis 8: Comparison: PF-04236921 50 mg vs Placebo; Week 8: Analysis was done using the ANCOVA model; CI parameter being the LS mean difference from that model; Test type: Superiority; LS mean difference = 3.93, 90% CI 2-sided [-2.75 to 10.62]
Statistical Analysis 9: Comparison: PF-04236921 50 mg vs Placebo; Week 12: Analysis was done using the ANCOVA model; CI parameter being the LS mean difference from that model; Test type: Superiority; LS mean difference = -0.78, 90% CI 2-sided [-7.47 to 5.91]
Statistical Analysis 10: Comparison: PF-04236921 50 mg vs Placebo; Week 16: Analysis was done using the ANCOVA model; CI parameter being the LS mean difference from that model; Test type: Superiority; LS mean difference = 3.67, 90% CI [-3.02 to 10.35]
Statistical Analysis 11: Comparison: PF-04236921 50 mg vs Placebo; Week 20: Analysis was done using the ANCOVA model; CI parameter being the LS mean difference from that model; Test type: Superiority; LS mean difference = 2.99, 90% CI 2-sided [-3.70 to 9.68]
Statistical Analysis 12: Comparison: PF-04236921 50 mg vs Placebo; Week 24: Analysis was done using the ANCOVA model; CI parameter being the LS mean difference from that model; Test type: Superiority; LS mean difference = 1.44, 90% CI 2-sided [-5.24 to 8.13]

22. Secondary Outcome: Change From Baseline in Short Form-6 Dimension (SF-6D) at Week 4, 8, 12, 16, 20 and 24
Description: The SF-6D focuses on seven of the eight health domains covered by the SF-36 Health Survey: physical functioning, role participation (combined role-physical and role-emotional), social functioning, bodily pain, mental health, and vitality. The SF-6D is an attempt to derive a single index from the SF-36 Health Survey for use in economic evaluation studies. As such, it represents a summary score based on a subset of the SF-36 data. Consequently, in lieu of the SF-6D, PCS and MCS SF-36 results are being provided. The score for each aspect and PCS/MCS is an average of the individual question scores, which are scaled 0-100 (100=highest level of functioning). LOCF method was used to impute missing values.
Time Frame: Baseline, Week 4, 8, 12, 16, 20, 24
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | PF-04236921 10 Milligram (10 mg) | PF-04236921 50 mg | Placebo
Number analyzed (Participants) | 45 | 47 | 45
Units on a scale
  MCS: Week 4: number analyzed (Participants) | 43 | 45 | 45
  MCS: Week 4 | 1.97 [-0.69 to 4.64] | 1.45 [-1.14 to 4.04] | 1.45 [-1.12 to 4.02]
  MCS: Week 8: number analyzed (Participants) | 43 | 46 | 45
  MCS: Week 8 | 1.57 [-1.10 to 4.23] | 1.97 [-0.59 to 4.52] | 2.05 [-0.52 to 4.62]
  MCS: Week 12: number analyzed (Participants) | 43 | 46 | 45
  MCS: Week 12 | 3.80 [1.13 to 6.46] | 2.50 [-0.06 to 5.05] | 2.52 [-0.05 to 5.09]
  MCS: Week 16: number analyzed (Participants) | 43 | 46 | 45
  MCS: Week 16 | 4.73 [2.07 to 7.40] | 2.79 [0.24 to 5.35] | 2.95 [0.38 to 5.52]
  MCS: Week 20: number analyzed (Participants) | 43 | 46 | 45
  MCS: Week 20 | 4.49 [1.82 to 7.15] | 1.71 [-0.85 to 4.26] | 3.28 [0.71 to 5.85]
  MCS: Week 24: number analyzed (Participants) | 43 | 46 | 45
  MCS: Week 24 | 2.94 [0.28 to 5.60] | 2.14 [-0.41 to 4.70] | 2.85 [0.28 to 5.42]
  PCS: Week 4: number analyzed (Participants) | 43 | 45 | 45
  PCS: Week 4 | 3.95 [1.75 to 6.15] | 3.24 [1.10 to 5.38] | 1.28 [-0.85 to 3.40]
  PCS: Week 8: number analyzed (Participants) | 43 | 46 | 45
  PCS: Week 8 | 5.48 [3.27 to 7.68] | 4.79 [2.68 to 6.90] | 2.11 [-0.01 to 4.23]
  PCS: Week 12: number analyzed (Participants) | 43 | 46 | 45
  PCS: Week 12 | 6.06 [3.86 to 8.26] | 4.66 [2.55 to 6.77] | 2.82 [0.70 to 4.95]
  PCS: Week 16: number analyzed (Participants) | 43 | 46 | 45
  PCS: Week 16 | 6.25 [4.05 to 8.45] | 4.50 [2.39 to 6.61] | 2.48 [0.36 to 4.60]
  PCS: Week 20: number analyzed (Participants) | 43 | 46 | 45
  PCS: Week 20 | 6.39 [4.19 to 8.59] | 5.63 [3.52 to 7.74] | 3.29 [1.17 to 5.42]
  PCS: Week 24: number analyzed (Participants) | 43 | 46 | 45
  PCS: Week 24 | 5.98 [3.77 to 8.18] | 5.53 [3.42 to 7.64] | 2.94 [0.82 to 5.06]
Statistical Analysis 1: Comparison: PF-04236921 10 Milligram (10 mg) vs Placebo; MCS Week 4: Analysis was done using the ANCOVA model; CI parameter being the LS mean difference from that model; Test type: Superiority; LS mean difference = 0.53, 90% CI 2-sided [-2.53 to 3.59]
Statistical Analysis 2: Comparison: PF-04236921 10 Milligram (10 mg) vs Placebo; MCS Week 8: Analysis was done using the ANCOVA model; CI parameter being the LS mean difference from that model; Test type: Superiority; LS mean difference = -0.48, 90% CI 2-sided [-3.54 to 2.58]
Statistical Analysis 3: Comparison: PF-04236921 10 Milligram (10 mg) vs Placebo; MCS Week 12: Analysis was done using the ANCOVA model; CI parameter being the LS mean difference from that model; Test type: Superiority; LS mean difference = 1.28, 90% CI 2-sided [-1.78 to 4.34]
Statistical Analysis 4: Comparison: PF-04236921 10 Milligram (10 mg) vs Placebo; MCS Week 16: Analysis was done using the ANCOVA model; CI parameter being the LS mean difference from that model; Test type: Superiority; LS mean difference = 1.78, 90% CI 2-sided [-1.28 to 4.84]
Statistical Analysis 5: Comparison: PF-04236921 10 Milligram (10 mg) vs Placebo; MCS Week 20: Analysis was done using the ANCOVA model; CI parameter being the LS mean difference from that model; Test type: Superiority; LS mean difference = 1.20, 90% CI 2-sided [-1.86 to 4.26]
Statistical Analysis 6: Comparison: PF-04236921 10 Milligram (10 mg) vs Placebo; MCS Week 24: Analysis was done using the ANCOVA model; CI parameter being the LS mean difference from that model; Test type: Superiority; LS mean difference = 0.09, 90% CI 2-sided [-2.98 to 3.15]
Statistical Analysis 7: Comparison: PF-04236921 50 mg vs Placebo; MCS Week 4: Analysis was done using the ANCOVA model; CI parameter being the LS mean difference from that model; Test type: Superiority; LS mean difference = 0.00, 90% CI 2-sided [-3.03 to 3.03]
Statistical Analysis 8: Comparison: PF-04236921 50 mg vs Placebo; MCS Week 8: Analysis was done using the ANCOVA model; CI parameter being the LS mean difference from that model; Test type: Superiority; LS mean difference = -0.09, 90% CI 2-sided [-3.09 to 2.92]
Statistical Analysis 9: Comparison: PF-04236921 50 mg vs Placebo; MCS Week 12: Analysis was done using the ANCOVA model; CI parameter being the LS mean difference from that model; Test type: Superiority; LS mean difference = -0.02, 90% CI 2-sided [-3.03 to 2.99]
Statistical Analysis 10: Comparison: PF-04236921 50 mg vs Placebo; MCS Week 16: Analysis was done using the ANCOVA model; CI parameter being the LS mean difference from that model; Test type: Superiority; LS mean difference = -0.16, 90% CI 2-sided [-3.17 to 2.85]
Statistical Analysis 11: Comparison: PF-04236921 50 mg vs Placebo; MCS Week 20: Analysis was done using the ANCOVA model; CI parameter being the LS mean difference from that model; Test type: Superiority; LS mean difference = -1.58, 90% CI 2-sided [-4.58 to 1.43]
Statistical Analysis 12: Comparison: PF-04236921 50 mg vs Placebo; MCS Week 24: Analysis was done using the ANCOVA model; CI parameter being the LS mean difference from that model; Test type: Superiority; LS mean difference = -0.71, 90% CI 2-sided [-3.72 to 2.30]
Statistical Analysis 13: Comparison: PF-04236921 10 Milligram (10 mg) vs Placebo; PCS Week 4: Analysis was done using the ANCOVA model; CI parameter being the LS mean difference from that model; Test type: Superiority; LS mean difference = 2.67, 90% CI 2-sided [0.14 to 5.20]
Statistical Analysis 14: Comparison: PF-04236921 10 Milligram (10 mg) vs Placebo; PCS Week 8: Analysis was done using the ANCOVA model; CI parameter being the LS mean difference from that model; Test type: Superiority; LS mean difference = 3.36, 90% CI 2-sided [0.84 to 5.89]
Statistical Analysis 15: Comparison: PF-04236921 10 Milligram (10 mg) vs Placebo; PCS Week 12: Analysis was done using the ANCOVA model; CI parameter being the LS mean difference from that model; Test type: Superiority; LS mean difference = 3.23, 90% CI 2-sided [0.70 to 5.76]
Statistical Analysis 16: Comparison: PF-04236921 10 Milligram (10 mg) vs Placebo; PCS Week 16: Analysis was done using the ANCOVA model; CI parameter being the LS mean difference from that model; Test type: Superiority; LS mean difference = 3.77, 90% CI 2-sided [1.24 to 6.30]
Statistical Analysis 17: Comparison: PF-04236921 10 Milligram (10 mg) vs Placebo; PCS Week 20: Analysis was done using the ANCOVA model; CI parameter being the LS mean difference from that model; Test type: Superiority; LS mean difference = 3.10, 90% CI 2-sided [0.57 to 5.63]
Statistical Analysis 18: Comparison: PF-04236921 10 Milligram (10 mg) vs Placebo; PCS Week 24: Analysis was done using the ANCOVA model; CI parameter being the LS mean difference from that model; Test type: Superiority; LS mean difference = 3.03, 90% CI [0.50 to 5.56]
Statistical Analysis 19: Comparison: PF-04236921 50 mg vs Placebo; PCS Week 4: Analysis was done using the ANCOVA model; CI parameter being the LS mean difference from that model; Test type: Superiority; LS mean difference = 1.96, 90% CI 2-sided [-0.53 to 4.46]
Statistical Analysis 20: Comparison: PF-04236921 50 mg vs Placebo; PCS Week 8: Analysis was done using the ANCOVA model; CI parameter being the LS mean difference from that model; Test type: Superiority; LS mean difference = 2.68, 90% CI [0.20 to 5.17]
Statistical Analysis 21: Comparison: PF-04236921 50 mg vs Placebo; PCS Week 12: Analysis was done using the ANCOVA model; CI parameter being the LS mean difference from that model; Test type: Superiority; LS mean difference = 1.84, 90% CI 2-sided [-0.65 to 4.32]
Statistical Analysis 22: Comparison: PF-04236921 50 mg vs Placebo; PCS Week 16: Analysis was done using the ANCOVA model; CI parameter being the LS mean difference from that model; Test type: Superiority; LS mean difference = 2.01, 90% CI 2-sided [-0.47 to 4.50]
Statistical Analysis 23: Comparison: PF-04236921 50 mg vs Placebo; PCS Week 20: Analysis was done using the ANCOVA model; CI parameter being the LS mean difference from that model; Test type: Superiority; LS mean difference = 2.34, 90% CI 2-sided [-0.15 to 4.82]
Statistical Analysis 24: Comparison: PF-04236921 50 mg vs Placebo; PCS Week 24: Analysis was done using the ANCOVA model; CI parameter being the LS mean difference from that model; Test type: Superiority; LS mean difference = 2.59, 90% CI 2-sided [0.11 to 5.08]

23. Secondary Outcome: Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F) Score at Baseline
Description: FACIT-F is a 13-item questionnaire. Participants scored each item on a 5-point scale: 0 (not at all) to 4 (very much). Larger the participant's response to the questions (with the exception of 2 negatively stated), greater was the participant's fatigue. For all questions, except for the 2 negatively stated ones, the code was reversed and a new score was calculated as (4 minus the participant's response). The sum of all responses resulted in the FACIT-Fatigue score for a total possible score of 0 (worse score) to 52 (better score).
Time Frame: Baseline
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | PF-04236921 10 Milligram (10 mg) | PF-04236921 50 mg | Placebo
Number analyzed (Participants) | 45 | 47 | 45
Units on a scale | 25.91 (1.700) | 29.38 (1.506) | 25.96 (1.760)

24. Secondary Outcome: Change From Baseline in Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F) Score at Week 4, 8, 12, 16, 20 and 24
Description: FACIT-F is a 13-item questionnaire. Participants scored each item on a 5-point scale: 0 (not at all) to 4 (very much). Larger the participant's response to the questions (with the exception of 2 negatively stated), greater was the participant's fatigue. For all questions, except for the 2 negatively stated ones, the code was reversed and a new score was calculated as (4 minus the participant's response). The sum of all responses resulted in the FACIT-Fatigue score for a total possible score of 0 (worse score) to 52 (better score). LOCF method was used to impute missing values.
Time Frame: Baseline, Week 4, 8, 12, 16, 20, 24
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | PF-04236921 10 Milligram (10 mg) | PF-04236921 50 mg | Placebo
Number analyzed (Participants) | 45 | 47 | 45
Units on a scale
  Week 4: number analyzed (Participants) | 43 | 45 | 45
  Week 4 | 3.16 [0.25 to 6.07] | 2.77 [-0.05 to 5.60] | 1.08 [-1.72 to 3.89]
  Week 8: number analyzed (Participants) | 43 | 46 | 45
  Week 8 | 4.39 [1.49 to 7.30] | 3.41 [0.62 to 6.20] | 2.44 [-0.37 to 5.24]
  Week 12: number analyzed (Participants) | 43 | 46 | 45
  Week 12 | 5.07 [2.16 to 7.97] | 3.59 [0.80 to 6.38] | 2.26 [-0.54 to 5.06]
  Week 16: number analyzed (Participants) | 43 | 46 | 45
  Week 16 | 5.81 [2.90 to 8.72] | 5.53 [2.74 to 8.32] | 1.93 [-0.88 to 4.73]
  Week 20: number analyzed (Participants) | 43 | 46 | 45
  Week 20 | 5.37 [2.46 to 8.28] | 4.32 [1.53 to 7.11] | 3.42 [0.61 to 6.22]
  Week 24: number analyzed (Participants) | 43 | 46 | 45
  Week 24 | 4.39 [1.49 to 7.30] | 3.30 [0.51 to 6.09] | 2.70 [-0.10 to 5.51]
Statistical Analysis 1: Comparison: PF-04236921 10 Milligram (10 mg) vs Placebo; Week 4: Analysis was done using the ANCOVA model; CI parameter being the Least Square (LS) mean difference from that model; Test type: Superiority; LS mean difference = 2.08, 90% CI 2-sided [-1.26 to 5.42]
Statistical Analysis 2: Comparison: PF-04236921 10 Milligram (10 mg) vs Placebo; Week 8: Analysis was done using the ANCOVA model; CI parameter being the LS mean difference from that model; Test type: Superiority; LS mean difference = 1.95, 90% CI 2-sided [-1.38 to 5.29]
Statistical Analysis 3: Comparison: PF-04236921 10 Milligram (10 mg) vs Placebo; Week 12: Analysis was done using the ANCOVA model; CI parameter being the LS mean difference from that model; Test type: Superiority; LS mean difference = 2.81, 90% CI 2-sided [-0.53 to 6.15]
Statistical Analysis 4: Comparison: PF-04236921 10 Milligram (10 mg) vs Placebo; Week 16: Analysis was done using the ANCOVA model; CI parameter being the LS mean difference from that model; Test type: Superiority; LS mean difference = 3.88, 90% CI 2-sided [0.54 to 7.22]
Statistical Analysis 5: Comparison: PF-04236921 10 Milligram (10 mg) vs Placebo; Week 20: Analysis was done using the ANCOVA model; CI parameter being the LS mean difference from that model; Test type: Superiority; LS mean difference = 1.95, 90% CI 2-sided [-1.39 to 5.29]
Statistical Analysis 6: Comparison: PF-04236921 10 Milligram (10 mg) vs Placebo; Week 24: Analysis was done using the ANCOVA model; CI parameter being the LS mean difference from that model; Test type: Superiority; LS mean difference = 1.69, 90% CI 2-sided [-1.65 to 5.03]
Statistical Analysis 7: Comparison: PF-04236921 50 mg vs Placebo; Week 4: Analysis was done using the ANCOVA model; CI parameter being the LS mean difference from that model; Test type: Superiority; LS mean difference = 1.69, 90% CI 2-sided [-1.61 to 4.99]
Statistical Analysis 8: Comparison: PF-04236921 50 mg vs Placebo; Week 8: Analysis was done using the ANCOVA model; CI parameter being the LS mean difference from that model; Test type: Superiority; LS mean difference = 0.97, 90% CI 2-sided [-2.31 to 4.26]
Statistical Analysis 9: Comparison: PF-04236921 50 mg vs Placebo; Week 12: Analysis was done using the ANCOVA model; CI parameter being the LS mean difference from that model; Test type: Superiority; LS mean difference = 1.33, 90% CI 2-sided [-1.96 to 4.61]
Statistical Analysis 10: Comparison: PF-04236921 50 mg vs Placebo; Week 16: Analysis was done using the ANCOVA model; CI parameter being the LS mean difference from that model; Test type: Superiority; LS mean difference = 3.60, 90% CI 2-sided [0.32 to 6.89]
Statistical Analysis 11: Comparison: PF-04236921 50 mg vs Placebo; Week 20: Analysis was done using the ANCOVA model; CI parameter being the LS mean difference from that model; Test type: Superiority; LS mean difference = 0.91, 90% CI 2-sided [-2.38 to 4.19]
Statistical Analysis 12: Comparison: PF-04236921 50 mg vs Placebo; Week 24: Analysis was done using the ANCOVA model; CI parameter being the LS mean difference from that model; Test type: Superiority; LS mean difference = 0.60, 90% CI 2-sided [-2.68 to 3.88]

ADVERSE EVENTS:
Description: An AE may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study. SAEs consist of all the SAEs including infectious SAEs; non-SAEs consist of all the non-SAEs including infectious non-SAEs.
Arm/Group | PF-04236921 10 Milligram (10 mg) | PF-04236921 50 mg | PF-04236921 200 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 4/45 | 3/47 | 7/46 | 8/45
Other Adverse Events (participants affected / at risk) | 20/45 | 24/47 | 32/46 | 26/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-04236921 10 Milligram (10 mg) (N=45) | PF-04236921 50 mg (N=47) | PF-04236921 200 mg (N=46) | Placebo (N=45)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 1
Cardio (Cardiac disorders) | 0 | 0 | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 1 | 0
Pericarditis (Cardiac disorders) | 0 | 0 | 1 | 1
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Metrorrhagia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Ovarian haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Umbilical hernia, obstructive (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Headache (Nervous system disorders) | 0 | 0 | 1 | 0
Vasculitis cerebral (Nervous system disorders) | 0 | 0 | 0 | 1
Aortic stenosis (Vascular disorders) | 0 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Visual impairment (Eye disorders) | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0
Arthroscopy (Investigations) | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Knee arthroplasty (Surgical and medical procedures) | 0 | 0 | 0 | 1
Acute sinusitis (Infections and infestations) | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1
Bronchopneumonia (Infections and infestations) | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 1
Disseminated tuberculosis (Infections and infestations) | 0 | 0 | 1 | 0
Infectious mononucleosis (Infections and infestations) | 1 | 0 | 0 | 0
Latent tuberculosis (Infections and infestations) | 0 | 0 | 0 | 1
Localised infection (Infections and infestations) | 1 | 0 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 0 | 1
Pyelonephritis chronic (Infections and infestations) | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PF-04236921 10 Milligram (10 mg) (N=45) | PF-04236921 50 mg (N=47) | PF-04236921 200 mg (N=46) | Placebo (N=45)
Abdominal pain (Gastrointestinal disorders) | 2 | 3 | 2 | 1
Abdominal pain upper (Gastrointestinal disorders) | 3 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 3 | 5 | 5
Nausea (Gastrointestinal disorders) | 3 | 4 | 6 | 7
Vomiting (Gastrointestinal disorders) | 1 | 2 | 2 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 4 | 3 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 3 | 3 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 4 | 2
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 3 | 5 | 2 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 1 | 3 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 3
Rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 4 | 1
Dizziness (Nervous system disorders) | 1 | 3 | 2 | 2
Headache (Nervous system disorders) | 4 | 8 | 5 | 2
Injection site pain (General disorders) | 0 | 3 | 2 | 1
Pyrexia (General disorders) | 0 | 2 | 0 | 3
Hepatic enzyme increased (Investigations) | 0 | 0 | 3 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 4 | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 0 | 2 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 3 | 3 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 3
Contusion (Injury, poisoning and procedural complications) | 3 | 1 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 1 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 4 | 2
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 3 | 0
Hypertension (Vascular disorders) | 4 | 2 | 4 | 1
Insomnia (Psychiatric disorders) | 1 | 1 | 3 | 2
Nephrolithiasis (Renal and urinary disorders) | 0 | 3 | 0 | 1
Bronchitis (Infections and infestations) | 5 | 6 | 3 | 3
Gastroenteritis (Infections and infestations) | 1 | 3 | 2 | 3
Pharyngitis (Infections and infestations) | 2 | 3 | 2 | 4
Sinusitis (Infections and infestations) | 1 | 3 | 4 | 0
Upper respiratory tract infection (Infections and infestations) | 5 | 6 | 11 | 7
Urinary tract infection (Infections and infestations) | 8 | 5 | 3 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.